CLINICAL TRIAL: NCT01191892
Title: A Randomized Phase II Trial of Carboplatin and Gemcitabine +/- Vandetanib in First Line Treatment of Advanced Urothelial Cell Cancer in Patients Who Are Not Suitable to Receive Cisplatin
Brief Title: Carboplatin and Gemcitabine Hydrochloride With or Without Vandetanib as First-Line Therapy in Treating Patients With Locally Advanced or Metastatic Urinary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000684016; WCTU-TOUCAN; ISRCTN-68146831; EUDRACT-2009-010140-33; EU-21066; CRUK-09/024; WCTU-SPON-672-09; ZENECA-WCTU-TOUCAN
Record Dates: First submitted 2010-08-29; First posted 2010-08-31 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Ureter Cancer; Urethral Cancer
Keywords: metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; transitional cell carcinoma of the bladder; stage III bladder cancer; stage IV bladder cancer; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; ureter cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — Carboplatin; Gemcitabine; vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Carboplatin, Gemcitabine and Placebo
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Drug: Placebo
- vandetanib (Experimental): Carboplatin, Gemcitabine and vandetanib
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Drug: vandetanib

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine hydrochloride
Drug: vandetanib
  Arms: vandetanib
Drug: Placebo — Placebo of vandetanib tablet
  Arms: Placebo

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vandetanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether giving carboplatin and gemcitabine hydrochloride is more effective with or without vandetanib as first-line therapy in treating urinary tract cancer.

PURPOSE: This randomized phase II trial is studying giving carboplatin together with gemcitabine hydrochloride and to see how well it works when given with or without vandetanib as first-line therapy in treating patients with locally advanced or metastatic urinary tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the antitumor activity (as measured by progression-free survival) of carboplatin and gemcitabine hydrochloride with versus without vandetanib as first-line treatment in patients with locally advanced or metastatic urothelial cell cancer who are not suitable to receive cisplatin.

Secondary

* To determine the safety, feasibility, and tolerability of these regimens in these patients.
* To determine the objective response rate.
* To determine the overall survival of patients treated with these regimens
* To assess the change of size of measurable lesions at 9 weeks of study therapy.

OUTLINE: This is a multicenter study. Patients are stratified according to relevant factors. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive carboplatin IV over 30 minutes on day 1, gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and an oral placebo once daily on days 1-21. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patient receive carboplatin and gemcitabine hydrochloride as in arm I. Patients also receive oral vandetanib once daily on days 1-21. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Blood and urine samples may be collected for laboratory analysis at baseline and after completion of study.

After completion of study treatment, patients are followed up at weeks 18, 26, 39, and 52.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma (pure or mixed histology) of the urothelium (upper or lower urinary tract)

  * Cancers with other pathologies are permitted provided the dominant morphology is transitional cell carcinoma
* Radiologically measurable disease according to RECIST v 1.1 criteria
* Locally advanced and/or metastatic disease not amenable to curative treatment with surgery or radiotherapy
* Patient not suitable for cisplatin therapy, meeting 1 or more of the following criteria:

  * More than 75 years of age
  * ECOG performance status > 2
  * Creatinine clearance < 30 mL/min
  * Clinically significant ischemic heart disease (myocardial infarction or unstable angina more than 3 but less than 12 months prior to date of randomization, symptomatic angina, or NYHA class I within 3 months prior to date of randomization)
  * Prior intolerance of cisplatin
  * Any other factor that, in the opinion of the investigator, indicates that cisplatin is not suitable for the patient (e.g., unilateral hearing loss)

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* ECOG performance status 0-2
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Creatinine clearance ≥ 30 mL/min
* Potassium ≥ 4.0 mmol/L OR below the CTCAE grade 1 upper limit
* Magnesium normal OR below the CTCAE grade 1 upper limit
* Serum calcium ≤ 2.9 mmol/L (If serum calcium is < lower limit of normal [LLN], then adjusted serum calcium must be ≥ LLN)
* ALT/AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN (< 5 times ULN if judged by the investigator to be related to liver metastases)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier-method contraception during and for 3 months (women) or 2 months (men) after completion of study therapy
* No evidence of severe or uncontrolled systemic disease or any concurrent condition that, in the investigator's opinion, makes it undesirable for the patient to participate in the trial or that would jeopardize compliance with the protocol
* No significant risk of cardiac complications, defined as any of the following:

  * Clinically significant cardiovascular event (e.g., myocardial infarction, superior vena cava syndrome [SVC], NYHA classification of heart disease ≥ class II within 3 months prior to entry, or presence of cardiac disease that, in the opinion of the investigator, significantly increases the risk of ventricular arrhythmia)
  * History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia

    * Atrial fibrillation, controlled on medication, is not exclusionary
* No QTc prolongation with other medications that requires discontinuation of that medication
* No congenital long QT syndrome or first-degree relative with unexplained sudden death under 40 years of age
* No QTc that is immeasurable or ≥ 480 msec on screening ECG

  * If a patient has a QTc interval ≥ 480 msec on screening ECG, the ECG screen may be repeated twice (at least 24 hours apart) and the average QTc from the three screening ECGs must be < 480 msec in order for the patient to be eligible for the study
  * Patients who are receiving a drug that has a risk of Torsades de Pointes are excluded if QTc is ≥ 460 msec
* No presence of left bundle branch block
* No hypertension not controlled by medical therapy (systolic blood pressure > 160 mm Hg or diastolic blood pressure > 100 mm Hg)
* No currently active diarrhea that, in the investigator's opinion, may affect the ability of the patient to either absorb vandetanib or to tolerate additional diarrhea episodes
* No previous or current malignancies of other histology within the past 5 years except for carcinoma in situ of the cervix, adequately treated basal cell or squamous cell carcinoma of the skin, or prostate cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior and no concurrent known potent CYP3A4 inducers (e.g., barbiturates, rifampicin, rifabutin, phenytoin, carbamazepine, troglitazone, phenobarbital, or St. John wort) or medication that has known adverse interactions with vandetanib

  * Dexamethasone (or equivalent) allowed as a pre-medication for chemotherapy
* At least 4 weeks since prior major surgery and complete surgical wound healing
* At least 30 days since prior and no other concurrent investigational agents
* No prior chemotherapy (unless delivered perioperatively and completed > 12 months prior to first presentation of recurrent disease)
* No other concurrent anticancer drug

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-06; Primary Completion 2015-12 (Actual); Study Completion 2016-09-05 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  Time to event PFS, follow-up to 1 year

SECONDARY OUTCOMES:
Tolerability and feasibility | 1 year
  Rate of randomisation and safety profile of randomised patients
Objective response rate as assessed by RECIST criteria | Up to 1 year
  Proportion of patients responding to treatment
Overall survival | 2 years
  Patients will be followed up until death by using NHS flagging service.
Change in size of measurable lesions 9 weeks after start of chemotherapy | 9 weeks
Toxicity during and after treatment as assessed by NCI CTCAE v 4.0 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jones, MD, Principal Investigator — University of Glasgow
Locations (21):
- United Kingdom (21):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Wales Cancer Trials Unit, Cardiff, Wales
  - Ayr Hospital, Ayr
  - Royal Bournemouth General Hospital, Bournemouth
  - Queens Hospital, Burton-on-Trent
  - Velindre Hospital, City and County of Cardiff
  - Western General Hospital, Edinburgh
  - Calderdale Royal Infirmary, Halifax
  - Huddersfield Royal Infirmary, Huddersfield
  - The Royal Lancaster Infirmary, Lancaster
  - St. James's University Hospital, Leeds
  - The Royal Free Hospital, London
  - St Marys Hospital, London
  - Charing Cross Hospital, London
  - Christie Hospital, Manchester
  - Mount Vernon Hospital, Northwood Middlesex
  - Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Surrey County Hospital, Surrey
  - The Royal Marsden Hospital, Surrey